CLINICAL TRIAL: NCT00852098
Title: Randomized Clinic Trial of Total Fundoplication and Fundal Mobilization With or Without Division of Short Gastric Vessels: Long-Term Endoscopic Evaluation
Brief Title: Laparoscopic Nissen Fundoplication Comparing Division Versus Non-Division of Short Gastric Vessels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of São Paulo (Other)
Collaborators: Hospital State Public (Unknown)
Responsible Party: JOSÉ FRANCISCO DE MATTOS FARAH, FEDERAL UNIVERSITY OF SÃO PAULO
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1069/06
Record Dates: First submitted 2009-02-25; First posted 2009-02-26 (Estimated); Last update posted 2009-02-26 (Estimated); Status verified 2009-02

CONDITIONS: Gastroesophageal Reflux
Keywords: Fundoplication; gastroesophageal reflux; gastric vessels; surgery
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Fundoplication; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): dividing short gastric vessels
  Interventions: Procedure: Lap Nissen fundoplication with division of short gastric vessels
- 2 (Active Comparator): non-dividing short gastric vessels
  Interventions: Procedure: Laparoscopic Nissen fundoplication without division of short gastric vessels

INTERVENTIONS:
Procedure: Lap Nissen fundoplication with division of short gastric vessels — Dividing short gastric vessels
  Other Names: Fundoplication, Gastroesophageal Reflux,Surgery
  Arms: 1
Procedure: Laparoscopic Nissen fundoplication without division of short gastric vessels — non-dividing short gastric vessels
  Other Names: Fundoplication, Gastroesophageal Reflux,Surgery
  Arms: 2

SUMMARY:
Recently, total fundoplication followed by laparoscopic esophageal hiatoplasty has been the most common surgical treatment for gastro-esophageal reflux. Although this procedure is effective, some patients still develop complications. Indeed, dividing the short gastric vessels is claimed by many authors to confer benefit to patients even it could not be proved in other studies. In an attempt to evaluate the role of dividing the short gastric vessels and its long-term impact on the surgical treatment of the gastro-esophageal reflux, the investigators initiated a randomized clinical trial to clarify this important fact. Patients were recruited for this trial and short-term results had been already published in a national journal. The investigators are now registering this study which particularly focuses on the endoscopic outcome evaluated on long-term basis after gastro-esophageal reflux surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

* objective gastroesophageal reflux in adults

Exclusion Criteria:

* esophageal motility disorder
* hard stenosis
* previous antireflux surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 1997-11; Primary Completion 2000-01 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Evaluate outcomes after Laparoscopic Nissen comparing division and non-division of short gastric vessels. | two years

SECONDARY OUTCOMES:
Long-term clinical and endoscopic outcome | 8-10 years

CONTACTS AND LOCATIONS:
Overall Officials: José Carlos DelGrande, MD, Study Director — Federal University of São Paulo; Michelle L DeOliveira, MD, Study Chair — Federal University of São Paulo; Francisco Farah, MD, Principal Investigator — Federal University of São Paulo; Renato Lupinacci, MD, Study Chair — Hospital State Public Server São Paulo
Locations (2):
- Brazil (2):
  - Federal University of São Paulo - UNIFESP, São Paulo, São Paulo
  - State Public Server of São Paulo Hospital (HSPE), São Paulo, São Paulo

REFERENCES:
- [Background] Yang H, Watson DI, Lally CJ, Devitt PG, Game PA, Jamieson GG. Randomized trial of division versus nondivision of the short gastric vessels during laparoscopic Nissen fundoplication: 10-year outcomes. Ann Surg. 2008 Jan;247(1):38-42. doi: 10.1097/SLA.0b013e31814a693e. PMID 18156921
- [Background] O'Boyle CJ, Watson DI, Jamieson GG, Myers JC, Game PA, Devitt PG. Division of short gastric vessels at laparoscopic nissen fundoplication: a prospective double-blind randomized trial with 5-year follow-up. Ann Surg. 2002 Feb;235(2):165-70. doi: 10.1097/00000658-200202000-00001. PMID 11807353
- [Background] Watson DI, Jamieson GG, Lally C, Archer S, Bessell JR, Booth M, Cade R, Cullingford G, Devitt PG, Fletcher DR, Hurley J, Kiroff G, Martin CJ, Martin IJ, Nathanson LK, Windsor JA; International Society for Diseases of the Esophagus--Australasian Section. Multicenter, prospective, double-blind, randomized trial of laparoscopic nissen vs anterior 90 degrees partial fundoplication. Arch Surg. 2004 Nov;139(11):1160-7. doi: 10.1001/archsurg.139.11.1160. PMID 15545560
- [Result] Farah JF, Grande JC, Goldenberg A, Martinez JC, Lupinacci RA, Matone J. Randomized trial of total fundoplication and fundal mobilization with or without division of short gastric vessels: a short-term clinical evaluation. Acta Cir Bras. 2007 Nov-Dec;22(6):422-9. doi: 10.1590/s0102-86502007000600002. PMID 18235928
- See also: Related Info — http://www.umm.edu/general_surgery/nissen_fundo.htm